CLINICAL TRIAL: NCT04681625
Title: Randomised Intervention Multicentre Study to Evaluate the Effect of Pelvic Floor Muscle Training in Men With BPH and OAB Treated With Silodosin - The SILODOSING Study
Brief Title: Evaluation of Silodosin and Pelvic Floor Muscle Training in Men With Benign Prostatic Hyperplasia and Overactive Bladder
Acronym: SILODOSING
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Comenius University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 09072020
Record Dates: First submitted 2020-12-16; First posted 2020-12-23 (Actual); Last update posted 2023-12-07 (Actual); Status verified 2023-12

CONDITIONS: Benign Prostatic Hyperplasia (BPH); Overactive Bladder
Keywords: Benign prostatic hyperplasia; overactive bladder; silodosin; pelvic floor muscle training
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Bladder, Overactive

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard silodosin treatment (Active Comparator): Peroral treatment with silodosin at a dose of 8 mg daily
  Interventions: Behavioral: Pelvic floor muscle training (PFMT) with suppressive urgency technique
- Standard silodosin treatment with PFMT (Experimental): Peroral treatment with silodosin at a dose of 8 mg daily Intervention: Behavioural: Pelvic floor muscle training (PFMT) with suppressive urgency technique
  Interventions: Behavioral: Pelvic floor muscle training (PFMT) with suppressive urgency technique

INTERVENTIONS:
Behavioral: Pelvic floor muscle training (PFMT) with suppressive urgency technique — Pelvic floor muscle training with suppressive urgency technique:
  1. Education about proper urination training in the period without pathological urgency.
  2. Education about conscious urgency suppression through PFMT - suppressive urgency technique.
  3. Education on the principle and effect of PFMT.
  4. Exercises of varying intensity of pelvic floor muscles in different positions.
  5. Exercises to relax the pelvic floor muscles. Exercise 5 times a week for 20-30 minutes a day.

SUMMARY:
This study will evaluate the efficacy of pelvic floor muscle training in men with benign prostatic hyperplasia and overactive bladder treated with Silodosin.

DETAILED DESCRIPTION:
This is a randomised-intervention, parallel, multicentre study which will evaluate the efficacy of pelvic floor muscle training in men with benign prostatic hyperplasia and overactive bladder treated with silodosin.

ELIGIBILITY:
Inclusion criteria:

• willing to provide written informed consent

* men over 50 years with lower urinary tract symptoms and overactive bladder and benign prostatic hyperplasia
* persistence of overactive bladder despite 4 weeks of silodosin treatment
* symptoms of overactive bladder (urinary frequency and urgency with or without urinary incontinence) for ≥3 months prior to visit 1.
* willing and able to complete the 3-day voiding diary and questionnaires
* International Prostate Symptom Score (IPSS) score ≥8.
* experience an average of 8 or more micturition's per day over the 3-day diary period.
* experience an average of 2 episodes of urgency per day (grade 3 or 4) over the 3-diary period

Exclusion criteria:

* post-void residual volume (PVR) >200 mL
* evidence of Urinary Tract Infection and haematuria
* use anticholinergics, beta 3 mimetics within 4 weeks prior to Visit 1 and during the study
* oncological diseases of the lower urinary tract and prostate
* neurogenic bladder
* urethral strictures and bladder neck stenosis
* urolithiasis
* diabetes mellitus
* previous surgery of lower urinary tract
* stress urinary incontinence
* intermittent catheterisation
* chronic urinary tract infection
* previous botox treatment in the last 12 months
* chronic electrostimulation treatment of OAB in the last 12 months
* patient began or has changed a bladder training program or pelvic floor exercises less than 90 days before 1 visit
* cognitive deficits and dementia
* man has participated in an interventional trial within 30 days prior to Visit 1
* total daily urine production over 2500 mL according to voiding diary

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Men
Enrollment: 172 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Change in the number of voidings and intensity of urgencies during 24 hours using a micturition diary. | over 12 weeks of treatment
  The investigators will compare change in the number of voidings and the intensity of urgencies during 24 hours in the combined silodosin and pelvic floor muscle training to silodosin treatment alone.

SECONDARY OUTCOMES:
Change in lower urinary tract symptoms. | over 12 weeks of treatment
  To examine changes in the score of lower urinary tract symptoms (LUTS) by the International Prostate Symptom Score (IPSS) in the combined silodosin and pelvic floor muscle training to silodosin treatment alone. 0 = minimum score, 35 = maximum score.
Change in incontinence quality of life . | over 12 weeks of treatment
  To examine change in incontinence quality of life by Overactive Bladder Questionnaire (OAB - q) in the combined silodosin and pelvic floor muscle training to silodosin treatment alone.
  0 = the worst to 100 = the best quality of life.
Change in patient global impression of improvement | over 12 weeks of treatment
  To examine changes in patient global impression of improvement in the combined silodosin and pelvic floor muscle training to silodosin treatment alone . 1 = much better. 7 = definitely worse.
Incidence of adverse events . | over 12 weeks of treatment
  To examine the incidence of adverse events in the combined silodosin and pelvic floor muscle training to silodosin treatment alone.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Svihra, Prof,MD,PhD, Study Director — Department of Urology, Jessenius Faculty of Medicine, Comenius University Bratislava Slovak Republic; Magdalena Hagovska, Assoc.pr.PhD, Study Chair — Faculty of Medicine, PJ Safarik University, Kosice, Slovak Republic
Locations (1):
- Jan Svihra, Martin, Slovakia

IPD SHARING:
Plan to Share IPD: No